CLINICAL TRIAL: NCT03288428
Title: Analgesia Comparison of Nalbuphine and Morphine for Laparoscopic Myomectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Yan Zhou, MD, MD, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NABUMORPHINE
Record Dates: First submitted 2017-06-11; First posted 2017-09-20 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Nalbuphine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nalbuphine (Experimental): using nalbuphine for patient controlled analgesia
  Interventions: Drug: Nalbuphine
- morphine (Active Comparator): using morphine for patient controlled analgesia
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Nalbuphine — patient controlled analgesia with Nalbuphine
  Arms: nalbuphine
Drug: Morphine — patient controlled analgesia with Morphine
  Arms: morphine

SUMMARY:
to compare the analgesia and side effect of nalbuphine and morphine for elective Laparoscopic myomectomy.

DETAILED DESCRIPTION:
To compare the analgesia and side effect of nalbuphine and morphine for elective Laparoscopic myomectomy, by using patient controlled analgesia postoperatively, a randomized, double blind clinical trial. Patients undergoing elective Laparoscopic myomectomy are randomly divided into two groups: nalbuphine and morphine groups. All patients are under general anesthesia with routine methods. The nalbuphine group receive postoperative patient controlled analgesia using nalbuphine 30mg/120ml, while the morphine group receive postoperative patient controlled analgesia using morphine 60mg/120ml. Perioperative parameters are to be collected to compare the two groups.

ELIGIBILITY:
Inclusion Criteria:

* elective Laparoscopic myomectomy patients 24hr post-operative patient controlled analgesia analgesia no mild or severe liver or renal disfunction

Exclusion Criteria:

* can't understand patient controlled analgesia device refuse trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
numerical rating scale | 24 hr post-operatively
  1-10

CONTACTS AND LOCATIONS:
Locations (1):
- First hospital Peking University, Beijing, Beijing Municipality, China